CLINICAL TRIAL: NCT01978639
Title: Outcomes of Single Injections of FloGraft Therapy, Autologous Stem Cells, or Platelet Rich Plasma for the Treatment of Pain in the Lumbar Facet Joints, Sacroiliac Joints, Upper Extremity Joints, and Lower Extremity Joints
Brief Title: Injections of FloGraft Therapy, Autologous Stem Cells, or Platelet Rich Plasma for the Treatment of Degenerative Joint Pain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Arizona Pain Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: APS 2013-022; 2013-022 (Other: Scottsdale Healthcare IRB)
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will assess the outcomes of three currently available regenerative treatments (FloGraft, autologous stem cell therapy, platelet rich plasma therapy) for painful degenerative conditions of the joints. Patients receiving one these treatments will be assessed before the treatment procedure and followed up at four points over the six months after their procedure. Patients' pain, quality of life, and pain medication use at follow up will be compared to baseline levels. The investigators hypothesize that all three treatments will be effective in reducing pain, improving quality of life, and reducing pain medication usage.

DETAILED DESCRIPTION:
This is an open-label, non-randomized study assessing the efficacy of three potentially regenerative treatments for degenerative conditions of the joints of the lower back (facet, sacroiliac), upper extremities (e.g., shoulder), and lower extremities (e.g., hip, knee). These treatments are:

1. A single injection of Applied Biologics' FloGraftTM.
2. A single injection of autologous bone marrow derived stem cells.
3. A single injection of platelet rich plasma.

Subjects will be assessed prior to treatment for their level of pain, quality of life, and pain medication usage. Subjects will be followed up at 4 weeks, 8 weeks, 12 weeks, and 24 weeks after treatment. At each of these follow up visits, pain, quality of life, and pain medication usage will be assessed.

The investigators hypothesize that all three treatment groups will experience reduced pain, improved quality of life, and reduced pain medication usage at follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older,
* Ability to complete follow-up visits,
* Able to understand the study protocol and provide consent,
* Significant pain (average pain in the past month greater than or equal to 5, from 0-10),
* Pain lasting at least 3 months,
* Pain associated with one of the following conditions: lumbar facet degeneration, - OR -degenerative condition causing upper extremity joint pain, - OR - degenerative condition causing lower extremity joint pain.

Exclusion Criteria:

* Current litigation or worker's compensation claim,
* Unstable pain medication dosage,
* Previous surgery at the affected site,
* Injections at the affected site within the past 6 months,
* Uncontrolled psychiatric condition,
* Pregnancy or lactating in women,
* History of adverse reactions to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults age 18 or older
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | 24 week follow up
  Worst pain in the past 24 hours, from 0 (no pain) to 10 (pain as bad as you can imagine).

SECONDARY OUTCOMES:
Oswestry Disability Index | 24 week follow up
  Total score from the Oswestry Disability Index
SF-36 | 24 week follow up
  Total score from the SF-36
Pain Medications survey | 24 week follow up
  Reduction in reported pain medication usage.
Global Pain Scale | 24 week follow up
  Levels of pain, emotional health, quality of life, and activities of daily living.
Adverse Events | 24 week follow up
  Any adverse events between the study procedure and the 24 week follow up will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Tory McJunkin, MD, Principal Investigator — Arizona Pain Specialists
Locations (1):
- Arizona Pain Specialists, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mobasheri A, Csaki C, Clutterbuck AL, Rahmanzadeh M, Shakibaei M. Mesenchymal stem cells in connective tissue engineering and regenerative medicine: applications in cartilage repair and osteoarthritis therapy. Histol Histopathol. 2009 Mar;24(3):347-66. doi: 10.14670/HH-24.347. PMID 19130405
- [Background] Diaz-Prado S, Rendal-Vazquez ME, Muinos-Lopez E, Hermida-Gomez T, Rodriguez-Cabarcos M, Fuentes-Boquete I, de Toro FJ, Blanco FJ. Potential use of the human amniotic membrane as a scaffold in human articular cartilage repair. Cell Tissue Bank. 2010 May;11(2):183-95. doi: 10.1007/s10561-009-9144-1. Epub 2010 Apr 13. PMID 20386989
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Lee KB, Hui JH, Song IC, Ardany L, Lee EH. Injectable mesenchymal stem cell therapy for large cartilage defects--a porcine model. Stem Cells. 2007 Nov;25(11):2964-71. doi: 10.1634/stemcells.2006-0311. Epub 2007 Jul 26. PMID 17656639
- [Background] Wakitani S, Imoto K, Yamamoto T, Saito M, Murata N, Yoneda M. Human autologous culture expanded bone marrow mesenchymal cell transplantation for repair of cartilage defects in osteoarthritic knees. Osteoarthritis Cartilage. 2002 Mar;10(3):199-206. doi: 10.1053/joca.2001.0504. PMID 11869080
- [Background] Sampson S, Reed M, Silvers H, Meng M, Mandelbaum B. Injection of platelet-rich plasma in patients with primary and secondary knee osteoarthritis: a pilot study. Am J Phys Med Rehabil. 2010 Dec;89(12):961-9. doi: 10.1097/PHM.0b013e3181fc7edf. PMID 21403592
- [Background] Filardo G, Kon E, Buda R, Timoncini A, Di Martino A, Cenacchi A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular knee injections for the treatment of degenerative cartilage lesions and osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2011 Apr;19(4):528-35. doi: 10.1007/s00167-010-1238-6. Epub 2010 Aug 26. PMID 20740273